CLINICAL TRIAL: NCT03045094
Title: Neck Flexion and Extension Implicate the Tracheal Tube-tip Displacement in Children Undergoing Head and Neck Surgeries
Brief Title: Neck Movement Implicate the Tracheal Tube-tip Displacement in Pediatric Surgery
Status: Completed | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Yan Siyi, Attending Doctor, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: 12015C1043
Record Dates: First submitted 2017-02-01; First posted 2017-02-07 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Pediatric Anesthesia; Tracheal Intubation
Keywords: pediatric; intubation; neck movement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the effect of head and neck movement in children on endotracheal tube (ETT) tip displacement undergoing head-and-neck surgeries. The tube-tip displacement will be measured using flexible fiberoptic bronchoscope.

DETAILED DESCRIPTION:
In clinical application, especially in head-and-neck surgeries, the operators often change the position of children's head-neck for easy operating. Flexing the head resulted in the ETT moving towards the carina, and extension resulted in the tube being displaced in the opposite direction. Head and neck movement change the length of trachea as well: extending the head resulted in the extension of trachea, while flexing resulted in the opposite. Serious complications following from head and neck movement, such as accidental extubation and endobronchial intubation, threat children's life.

In pediatric anesthesia, insertion depth (cm) of orotracheal intubation equals to age/2+12, according to classic intubation formulae. The ETT will be put in the depth calculated by the classic formulae under general anesthesia. The distance of ETT-tip displacement and the length change of trachea will be measured as the head and neck placed as follows: fully extended, neutral position, or fully flexed. These three head and neck positions imitate the head-neck movement during those head-and-neck surgeries.

ELIGIBILITY:
Inclusion Criteria:

* subject has elective head-and-neck surgery schedule
* subject will have orotracheal intubation under general anesthesia

Exclusion Criteria:

* subject has malformations of the trachea or bronchus on chest X-ray
* subject has spinal deformity
* subject has difficulties in neck flexion or extension
* subject has neck pain

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who schedul to undergo elective head-and-neck surgeries under general anesthesia with orotracheal intubation will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Distance of trachea carina (TC) to endotracheal tube (ETT) tip | 10min (time that the measurement need)
  Measure the distance between trachea carina to the tip of ETT in three different neck-head positions: fully flexion, neutral positon and fully extension.

SECONDARY OUTCOMES:
Distance of tracheal length | 10min (time that the measurement need)
  Tracheal length equals the distance between trachea carina (TC) to posterior vocal commissure. Measure Tracheal length in three different neck-head positions: fully flexion, neutral positon and fully extension.
Serious complication of unexpected displacement of the endotracheal tube: accidental extubation | intraoperative
  When the operator put the child's neck into extension position, accidental extubation may occur, which can lead to hypoxia and asphyxia.
Serious complication of unexpected displacement of the endotracheal tube: endobronchial intubation. | intraoperative
  When the operator put the child's neck into flexion position, accidental endobronchial intubation may occur, which can lead to one-lung ventilation and pulmonary edema.

CONTACTS AND LOCATIONS:
Overall Officials: SIYI YAN, MD, Principal Investigator — Beijing Tsinghua Chang Gung Hospital
Locations (1):
- Department of Anesthesia, Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
After recruiting, upload the distance of trachea carina(TC) to endotracheal tube (ETT) tip and the distance of tracheal length of each volunteer.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Real time access

REFERENCES:
- [Background] Dronen S, Chadwick O, Nowak R. Endotracheal tip position in the arrested patient. Ann Emerg Med. 1982 Feb;11(2):116-7. doi: 10.1016/s0196-0644(82)80328-4. No abstract available. PMID 7137685
- [Background] McCoy EP, Russell WJ, Webb RK. Accidental bronchial intubation. An analysis of AIMS incident reports from 1988 to 1994 inclusive. Anaesthesia. 1997 Jan;52(1):24-31. doi: 10.1111/j.1365-2044.1997.007-az007.x. PMID 9014541
- [Background] Mariano ER, Ramamoorthy C, Chu LF, Chen M, Hammer GB. A comparison of three methods for estimating appropriate tracheal tube depth in children. Paediatr Anaesth. 2005 Oct;15(10):846-51. doi: 10.1111/j.1460-9592.2005.01577.x. PMID 16176312
- [Background] Lau N, Playfor SD, Rashid A, Dhanarass M. New formulae for predicting tracheal tube length. Paediatr Anaesth. 2006 Dec;16(12):1238-43. doi: 10.1111/j.1460-9592.2006.01982.x. PMID 17121553
- [Background] Gamble JJ, McKay WP, Wang AF, Yip KA, O'Brien JM, Plewes CE. Three-finger tracheal palpation to guide endotracheal tube depth in children. Paediatr Anaesth. 2014 Oct;24(10):1050-5. doi: 10.1111/pan.12452. Epub 2014 Jun 23. PMID 24958069
- [Background] Bloch EC, Ossey K, Ginsberg B. Tracheal intubation in children: a new method for assuring correct depth of tube placement. Anesth Analg. 1988 Jun;67(6):590-2. No abstract available. PMID 3377215
- [Background] Weiss M, Knirsch W, Kretschmar O, Dullenkopf A, Tomaske M, Balmer C, Stutz K, Gerber AC, Berger F. Tracheal tube-tip displacement in children during head-neck movement--a radiological assessment. Br J Anaesth. 2006 Apr;96(4):486-91. doi: 10.1093/bja/ael014. Epub 2006 Feb 7. PMID 16464981
- [Background] Jin-Hee K, Ro YJ, Seong-Won M, Chong-Soo K, Seong-Deok K, Lee JH, Jae-Hyon B. Elongation of the trachea during neck extension in children: implications of the safety of endotracheal tubes. Anesth Analg. 2005 Oct;101(4):974-977. doi: 10.1213/01.ane.0000169330.92707.1e. PMID 16192505
- [Background] Kim JT, Kim HJ, Ahn W, Kim HS, Bahk JH, Lee SC, Kim CS, Kim SD. Head rotation, flexion, and extension alter endotracheal tube position in adults and children. Can J Anaesth. 2009 Oct;56(10):751-6. doi: 10.1007/s12630-009-9158-y. Epub 2009 Jul 29. PMID 19639372